CLINICAL TRIAL: NCT05164289
Title: Interest of EMDR (Eye Movement Desensitization and Reprocessing) Psychotherapy in the Management of Schizophrenic Disorders
Brief Title: Interest of EMDR Schizophrenic Disorders
Acronym: EMDRpsychose
Status: Terminated | Type: Observational
Why Stopped: No patients included in the control group and inclusion rate too low.
Sponsor: Hôpital NOVO (Other)
Responsible Party: Sponsor
Other Study IDs: CHRD 1721
Record Dates: First submitted 2021-12-06; First posted 2021-12-20 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2022-05

CONDITIONS: Schizophrenic Disorders
Keywords: Schizophrenic disorders; Psychosis; Eye Movement Desensitization and Reprocessing
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Control Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Control group: Patients in the control group will have simple consultations on D15, D30, D45, D60 and D75
  Interventions: Other: Control group
- EMDR group: Patients in the EMDR group will have EMDR session on D15, D30, D45, D60 and D75
  Interventions: Other: EMDR group

INTERVENTIONS:
Other: Control group — Patients in the control group will have simple consultations on D15, D30, D45, D60 and D75
  Groups: Control group
Other: EMDR group — Patients in the EMDR group will have EMDR session on D15, D30, D45, D60 and D75
  Groups: EMDR group

SUMMARY:
The purpose of this study is to determine the interest of the use of EMDR (Eye Movement Desensitization and Reprocessing) psychotherapy in the management of psychotic disorders, in particular schizophrenic disorders.

DETAILED DESCRIPTION:
Since 2015 more and more studies conducted by researchers, especially Dutch and English, are interested in the use of EMDR (Eye Movement Desensitization and Reprocessing) for other pathologies such as bipolar disorder, unipolar depression, anxiety disorders, psychotic disorders, substance use disorders and chronic pain.

These studies show that EMDR appears to be a technique that is both effective, capable of significantly improving symptoms, and without risk for patients, while respecting the protocol and the clinical stabilization provided during the procedure.

To date, the use of EMDR for the management of psychotic patients has not been the subject of any prospective study in France and the authors' conclusions converge on the fact that it is essential to carry out more research on the subject.

For this, the investigators wish to evaluate the effect of EMDR on the management of patients with schizophrenic disorders, on the basis that this psychotherapy would improve their quality of life (improvement of all the specific scores used in psychiatry). : PANSS, DES, HAD and WEMWBS scales).

Finally, the investigators believe that it is relevant to assess the benefit of EMDR six months after hospitalization of patients, in order to measure the maintenance of this efficacy in the medium term

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years and over,
* Hospitalized for decompensated psychotic disorder, Positive diagnosis of schizophrenia or schizoaffective disorder (according to the DSM-V psychiatry manual),
* With positive or negative symptoms according to the Positive and Negative Syndrome Scale (PANSS),
* Stabilized clinical condition (considered compatible with hospital discharge),
* With ambulatory follow-up planned after hospitalization

Exclusion Criteria:

* < 18 years,
* Patients who do not meet the diagnostic criteria (according to the DSM-V psychiatry manual) for schizophrenic or schizoaffective disorder),
* Non-French speaking or illiterate patients,
* Cognitive disorders making it impossible the understanding and the none- opposition to the study,
* Non-stabilized clinical condition (incompatible with hospital discharge),

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized for decompensated psychotic disorder in the psychiatric departments of the Centers Hospitaliers of Pontoise or Villejuif.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2021-12-10 (Actual); Primary Completion 2022-04-27 (Actual); Study Completion 2022-04-27 (Actual)

PRIMARY OUTCOMES:
Assessment of the decrease in the severity of positive or negative symptoms of schizophrenia | At 6 month after Hospital discharge (M0)
  The decrease in the severity of positive or negative symptoms of schizophrenia is assessed using the "Positive and Negative Syndrome Scale" (PANSS) between M0 and M6.This decrease will be considered effective if it's greater than or equal to 20%.

SECONDARY OUTCOMES:
Assessment of the decrease in the intensity of dissociative symptoms. | At 6 month after Hospital discharge (M0)
  The decrease in the intensity of dissociative symptoms is assessed using the Dissociative Experience Scale (DES) between M0 and M6.
  The DES is a short written questionnaire. It consists of 28 items that assess the frequency of various dissociative symptoms in the patient's daily life.
  0 corresponds to the answer "Never" and 100 to the answer "All the time". The total score is obtained by adding the scores of the 28 items and then dividing by 28. This gives a score between 0 and 100.
Assessment of the decrease in the intensity of anxiety and depressive symptoms. | At 6 month after Hospital discharge (M0)
  The decrease in the intensity of anxiety and depressive symptoms is assessed using the Hospital Anxiety and Depression (HAD) between M0 and M6 The HAD scale is a short written questionnaire, consisting of 14 items to assess the patient's symptoms of anxiety and depression.
  The total anxiety score is obtained by adding the scores of items 1, 3, 5, 7, 9, 11 and 13 and the total depression score by adding the scores of the remaining items.
  The interpretation of the results is as follows:
  Score ≤ 7 = absence of symptomatology, 8 ≥ Score ≤ 10 = questionable symptomatology Score ≥ 11 = certain symptomatology.
Quality of life assessment | At 6 month after Hospital discharge (M0)
  The quality of life is assessed using the Warwick-Edinburgh Mental Well-Being Scale (WEMWBS).
  The Warwick-Edinburgh Mental Wellbeing Scale (WEMWBS) assesses the psychological well-being of individuals. It consists of 14 items on a likert scale of 5 (1: never, 2: rarely, 3: sometimes, 4: often, 5: all the time).
  In this scale, there is no threshold score, but the higher the score, the stronger the psychological well-being of the individual.
  An improvement in the quality of life is measured by an increase in the scale score between M0 and M6

CONTACTS AND LOCATIONS:
Overall Officials: Dr Marie-Claire ASMAR, Principal Investigator — Hospital René Dubos - Pontoise
Locations (2):
- France (2):
  - Departement of Psychiatry - Hospital René Dubos, Pontoise
  - Departement of Psychiatry -Hospital Paul Guiraud, Villejuif

IPD SHARING:
Plan to Share IPD: No